CLINICAL TRIAL: NCT06665126
Title: A Triple-Group Randomized Controlled Trial to Evaluate the Effects of a Prebiotic and Probiotic Supplement to Provide Relief From Symptoms Associated With Bacterial Vaginosis and Yeast Infections.
Brief Title: A Study to Evaluate the Effects of a Prebiotic and Probiotic Supplement to Provide Relief From Symptoms Associated With Bacterial Vaginosis and Yeast Infections.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Happy V (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20397
Record Dates: First submitted 2024-10-07; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Bacterial Vaginosis; Yeast Infection
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 3 groups (test product, active placebo, excipient placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blind design to ensure unbiased results. The three groups in the study (test product, active placebo, and excipient placebo) will receive capsules that are identical in appearance, taste, and packaging. Neither the participants, the investigators, nor the outcomes assessors will know which group the participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product Group (Experimental): Participants in this group will receive the test product, a prebiotic and probiotic supplement.
  Interventions: Dietary Supplement: Prebiotic + Probiotic Supplement
- Active Placebo Group (Placebo Comparator): Participants in this group will receive an active placebo.
  Interventions: Dietary Supplement: Active Placebo Supplement
- Excipient Placebo Group (Placebo Comparator): Participants in this group will receive an excipient placebo.
  Interventions: Dietary Supplement: Excipient Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Prebiotic + Probiotic Supplement — This intervention includes a combination of prebiotics and probiotics designed to promote vaginal and digestive health. The supplement contains Biotin, Lactobacillus acidophilus (as LA-14®), Bifidobacterium lactis (HN019™), Lactobacillus rhamnosus (as HN001™), Lactobacillus crispatus (as CCFM1110™), Lactobacillus gasseri (as HLG13™), Lactobacillus reuteri (as HR7™), Bacillus subtilis (as DE111®), PreforPro®, White Rice Flour, Magnesium Stearate (Vegetable Source), Silicon Dioxide (Bamboo Source), and Cellulose (Vegetable Capsule). Participants take two capsules daily with food for 30 days.
  Arms: Test Product Group
Dietary Supplement: Active Placebo Supplement — The active placebo supplement contains similar probiotic strains without the prebiotic component. Ingredients include Biotin, Lactobacillus acidophilus, Bifidobacterium lactis, Lactobacillus rhamnosus, Lactobacillus crispatus, Lactobacillus gasseri, Lactobacillus reuteri, Bacillus subtilis, Inulin (from Chicory Root), White Rice Flour, Magnesium Stearate (Vegetable Source), Silicon Dioxide (Bamboo Source), and Cellulose (Vegetable Capsule). Participants take two capsules daily with food for 30 days.
  Arms: Active Placebo Group
Dietary Supplement: Excipient Placebo Supplement — The excipient placebo supplement contains no active ingredients related to prebiotics or probiotics. It includes White Rice Flour, Magnesium Stearate (Vegetable Source), and Cellulose (Vegetable Capsule). Participants take two capsules daily with food for 30 days.
  Arms: Excipient Placebo Group

SUMMARY:
This virtual randomized controlled trial evaluates the efficacy of a prebiotic and probiotic supplement in providing relief from symptoms associated with bacterial vaginosis and yeast infections. Participants will be randomized into three groups-test product, active placebo, and excipient placebo-and will take two capsules daily for 30 days. The study will assess the effects on vaginal microbiome, symptoms of bacterial vaginosis and yeast infections, and overall vaginal health.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 25+
* Self-reported concerns symptoms associated with bacterial vaginosis or candida overgrowth, including itchiness, redness, abnormal discharge, and an unpleasant odor.
* Suffers from digestive issues, including bloating, gas, or other digestive discomfort.
* Generally healthy - do not live with any uncontrolled chronic diseases.
* Willing to avoid using any vaginal health-related medications, supplements, and herbal remedies for the duration of this study.
* If taking oral supplements or herbal remedies targeted at vaginal health, has been consistently taking these for at least 3 months prior to starting the study and is willing to maintain this routine for the study duration.

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Planning to undergo any procedure related to their vaginal health.
* Started any new medications or supplements that target vaginal health in the past 3 months.
* Anyone with known severe allergic reactions that require the use of an Epi-Pen, or any known allergies to any of the product ingredients
* Women who are pregnant, breastfeeding, or attempting to conceive
* Unwilling to follow the study protocol
* Anyone who has undergone any surgeries or invasive treatments in the last three months or has any planned during the study period.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Vaginal Microbiome | Baseline, Day 30
  This outcome measures the change in vaginal microbiome parameters from Baseline to Day 30. The vaginal microbiome will be assessed using microbiome sequencing at both Baseline and Day 30.

SECONDARY OUTCOMES:
Change in Perceived Symptoms of Bacterial Vaginosis | Baseline, Day 1, Day 7, Day 14, Day 21, Day 30
  This outcome measures the change in symptoms associated with bacterial vaginosis and yeast infections (e.g., itchiness, odor, abnormal discharge) as reported by participants through questionnaires.
Change in Perceived Symptoms of Yeast Infections | Baseline, Day 1, Day 7, Day 14, Day 21, Day 30
  This outcome measures the change in symptoms associated with bacterial vaginosis and yeast infections (e.g., itchiness, odor, abnormal discharge) as reported by participants through questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No